CLINICAL TRIAL: NCT02347215
Title: Changes in Ischemia and Angina Over One Year Among ISCHEMIA Trial Screen Failures
Brief Title: Changes in Ischemia and Angina Over 1 Year Among ISCHEMIA Trial Screen Failures With no Obstructive CAD on Coronary CT Angiography
Acronym: CIAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Duke Clinical Research Institute (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s11-00498
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Microvascular Angina; Angina Pectoris
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): All patients undergo quality of life assessment at 2-3 time points and stress imaging at two time points
  Interventions: Other: Quality of Life assessment; Procedure: Stress imaging

INTERVENTIONS:
Other: Quality of Life assessment — Seattle Angina Questionnaire and other questionnaires.
Procedure: Stress imaging — Stress imaging

SUMMARY:
Serial assessment of angina status and ischemia on stress echo over one year among patients with moderate ischemia on stress imaging and non-obstructive CAD on coronary CT angiography.

DETAILED DESCRIPTION:
Some people with chest pain are found to have open arteries on angiograms instead of blocked arteries and many, but not all, of these people have abnormal stress tests or other tests showing there is not enough blood flow to the heart. Prior research has not made clear whether chest pain in such patients is due to heart disease or something else, in part because no one has found out whether chest pain and stress test results change in the same direction over time. This study will use two measurements of chest pain and two stress tests, one year apart, to find out if chest pain and abnormal stress tests are both caused by the same problem: not enough blood flow to the heart.The association between angina, ischemia and atherosclerosis severity at baseline will be examined, as will medication effects.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled but not randomized in ISCHEMIA trial
* Stress echocardiography used for enrollment*
* No obstructive CAD on study coronary CT angiography (defined as no ≥50% stenosis in a major epicardial vessel)
* Ischemic symptoms (chest pain or other potential ischemic equivalent).
* Participant is willing to give written informed consent
* Age ≥ 21 years

Exclusion Criteria:

* Inability to comply with protocol
* Prior PCI or CABG

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) score | baseline-one year comparison

SECONDARY OUTCOMES:
Ischemia severity | baseline-one year comparison
Coronary atherosclerosis severity (comparison with SAQ score and with ischemia severity) | baseline
  comparison with SAQ score and with ischemia severity
Ischemia severity (comparison with SAQ score and with ischemia severity) | baseline
  comparison with SAQ score and with atherosclerosis severity
Medical therapy used for angina (comparison with SAQ score and ischemia severity) | one year
  comparison with SAQ score and ischemia severity
Major adverse cardiac events | one year
  death, MI, stroke, cardiovascular hospitalizations/ER visits

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hochman, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Medical Center and Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Hausvater A, Anthopolos R, Seltzer A, Spruill TM, Spertus JA, Peteiro J, Lopez-Sendon JL, Celutkiene J, Demchenko EA, Kedev S, Beleslin BD, Sidhu MS, Grodzinsky A, Fleg JL, Maron DJ, Hochman JS, Reynolds HR; CIAO-ISCHEMIA Research Group. Sex Differences in Psychosocial Factors and Angina in Patients With Chronic Coronary Disease. J Am Heart Assoc. 2025 Mar 4;14(5):e037909. doi: 10.1161/JAHA.124.037909. Epub 2025 Feb 25. PMID 39996455
- [Derived] Reynolds HR, Picard MH, Spertus JA, Peteiro J, Lopez Sendon JL, Senior R, El-Hajjar MC, Celutkiene J, Shapiro MD, Pellikka PA, Kunichoff DF, Anthopolos R, Alfakih K, Abdul-Nour K, Khouri M, Bershtein L, De Belder M, Poh KK, Beltrame JF, Min JK, Fleg JL, Li Y, Maron DJ, Hochman JS. Natural History of Patients With Ischemia and No Obstructive Coronary Artery Disease: The CIAO-ISCHEMIA Study. Circulation. 2021 Sep 28;144(13):1008-1023. doi: 10.1161/CIRCULATIONAHA.120.046791. Epub 2021 Jun 1. PMID 34058845